CLINICAL TRIAL: NCT01691027
Title: Visuomotor Rehabilitation Training for Manual Task Deficits From Macular Scotomas
Acronym: VRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1000-R
Record Dates: First submitted 2012-09-19; First posted 2012-09-24 (Estimated); Results first posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2017-08

CONDITIONS: Scotoma, Central; Central Visual Impairment
Keywords: scotoma, central; visual motor coordination
MeSH Terms: conditions — Scotoma; Blindness, Cortical

STUDY DESIGN:
Intervention Model Description: All eligible subjects trained on three computer-based training modules. SLO assessment of changes in fine manual task performance and in retinal functional geography was done before and after each training module.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Visuo-motor training for low vision (Experimental): All participants undergo training on scotoma awareness, Line and Circle Tracing and Video games
  Interventions: Behavioral: Visuo-motor training

INTERVENTIONS:
Behavioral: Visuo-motor training — Participants will undergo training on three developed software modules on Samsung Galaxy Note Pro tablets to see their effect on low vision rehabilitation
  Other Names: Scotoma Awareness; Line and Circle Tracing; Video games (Pong and PacMan)

SUMMARY:
The research is aimed at developing and testing a new method of visual-motor rehabilitation of Veterans with macular degeneration by using inexpensive "tablet" computers at home.

DETAILED DESCRIPTION:
The research objective is to test the hypothesis that practicing eye-hand coordination using tablet-computers can improve manual skills of those with Age-related Macular Degeneration (AMD). AMD causes the loss of sharp central vision used for reading and many other everyday activities. Those with AMD experience a "macular scotoma", a blanked-out area of whatever they're attempting to look at, and they must use an area of peripheral vision, the "Preferred Retinal Locus (PRL)" to look at objects of interest. The PRL does not provide sharp vision, causing deficits in eye-hand coordination needed for manual tasks. There have been few studies of visuo-motor rehabilitation training for deficits caused by macular scotomas. However, a recent study demonstrated that visuo-motor eye movement training dramatically improved reading ability of subjects with AMD. In addition, it has been shown that playing action video games can improve certain visual skills. Thus, a small but growing body of research suggests that it may be possible to ameliorate manual task deficits caused by AMD through computer-based visuo-motor rehabilitation training.

To test this idea, two visuo-motor training modules will be developed for low-cost tablet computers that subjects will use at home. Modules will be for, line and circle tracing, and video games. Both modules will involve PRL-hand coordination by moving a stylus on the tablet screen in response to stimuli. Line and circle tracing will develop eye-hand coordination skills needed for printing. The video game module will provide practice in PRL-hand coordination. Progress in PRL-hand coordination will be automatically recorded on the tablet-computer.

Changes in manual task performance from the training modules will be assessed after each training module using previously developed Scanning Laser Ophthalmoscope (SLO) tests of maze-tracing, and printing. The SLO will also be used to determine the position and fixation stability of the subject's PRL and the retinal position of the scotoma. SLO testing will be repeated three months after all training. Digitized SLO video images showing the hand, stylus, and object on the retina will be measured and analyzed. Several performance measures will be derived from the SLO image analysis including maze-tracing accuracy, printing legibility, retinal area of the stylus, percentage of time the stylus is in the scotoma, and PRL retinal area. This data will be statistically analyzed to determine whether visuo-motor training with the computer tablets improves manual task performance and whether one module is more effective than other.

There will be six groups of five subjects. Subjects will be assigned as they are recruited to a group until the group is full. Two groups will have training delayed by 6 months and will be tested on the SLO 4 times to assess changes in the dependent measure without training. Following training on each module, subject will be tested on maze tracing and printing in the SLO. Two groups undergo four SLO tests without training and begin training six months later.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral macular scotomas
* Preferred Retinal Locus (PRL) in at least one eye
* Visual acuity 20/400 or better in at least one eye
* No peripheral visual field loss
* No medications that could affect motor control
* Normal arm/hand range of motion
* Pass cognitive ability exam

Exclusion Criteria:

* No macular scotomas
* Visual acuity of 20/30 or better
* Medications that affect motor control
* Limited arm/hand range of motion
* Fail cognitive ability exam

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-07; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George T Timberlake, PhD, Principal Investigator — Kansas City VA Medical Center, Kansas City, MO
Locations (1):
- Kansas City VA Medical Center, Kansas City, MO, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with bilateral AMD, no foveal vision, and acuities poorer than 20/60 in each eye were screened in the eye clinic and those who met inclusion criteria were enrolled in the study. On each laboratory visit, subjects' eyes were checked for angle closure and, if angles wee open, dilated the eye to be tested
Pre-assignment Details: Enrolled subjects when found to have residual foveal vision in baseline SLO retinal functional map and/or are unable to follow the instructions for SLO testing were excluded from the study before training assignment.
Period: Scotoma Awareness
Arm/Group | Visuo-motor Training for Low Vision
Started | 4 (Four subjects started scotoma awareness training module)
Completed | 4 (Four subjects were able to complete scotoma awareness training module)
Not Completed | 0
Period: Line and Circle Tracing Training
Arm/Group | Visuo-motor Training for Low Vision
Started | 4 (Four subjects started line and circle tracing training module)
Completed | 4 (Four subjects were able to complete line and circle tracing training module.)
Not Completed | 0
Period: Video Games Training
Arm/Group | Visuo-motor Training for Low Vision
Started | 4 (Four subjects started video game training module)
Completed | 4 (Four subjects were able to complete video games training module)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: For each subject, SLO retinal functional maps are shown for Baseline, Pre-training, Post line and Circle Tracing training, and Post Video Game training for both maze tracing and printing. Tables show data derived from the retinal maps and associated performance measurement.
Groups:
- Crossover Design. All Subjects Undergo All Treatments.: Each participating subject will have three training modules on a tablet computer: scotoma awareness, line and curve tracing, and video games. The order of modules will be different for different groups of subjects. Training on a module will cease when the subject reaches a performance criterion. Retinal assessments will occur after each training module completion.
Arm/Group | Crossover Design. All Subjects Undergo All Treatments.
Number analyzed (Participants) | 4
Age, Continuous [Mean (Full Range); unit: Years] — Population: Only 4 subjects with ages in range of 65 to 92 participated and were able to complete all training.
  Years | 84.5 [65 to 92]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Four subjects 1 female and 3 males participated and completed all testing
  Participants
    Female | 1
    Male | 3
SLO retinal functional map [Mean (Full Range); unit: percent traced] | 80 [0 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Eye-hand Coordination
Description: Maze tracing represents the fine eye-hand coordination needed for a wide variety of manual tasks and an improvement in maze tracing indicates an improvement in eye-hand coordination
Time Frame: base line, pre-test, post tracing and videogames training
Population: Out of Ten selected subjects, 3 were rejected after completing Baseline SLO retinal function map because of residual foveal vision. Two subjects failed to follow the instructions for SLO testing. One subject completed initial phase but failed to complete testing because of medical problems. Four subjects were able to complete all testing.
Measure: Number; unit: Percentage
Groups:
- Visuo-motor Training: Participants undergo training on three modules, (1)scotoma awareness, (2) line and curve tracing, and (3) video games. SLO assessments of changes in fine manual task performance was measured by an improvement in mean maze tracing and printing score. Improvement in visuo-motor control was measured by stylus ellipse area and stylus-PRL distance before and after training.
Arm/Group | Visuo-motor Training
Number analyzed (Participants) | 4
Percentage
  Participant 1 baseline: number analyzed (Participants) | 1
  Participant 1 baseline | 42.8
  Participant 1 pretest: number analyzed (Participants) | 1
  Participant 1 pretest | 45.4
  Participant 1 post tracing: number analyzed (Participants) | 1
  Participant 1 post tracing | 30.4
  Participant 1 post gaming: number analyzed (Participants) | 1
  Participant 1 post gaming | 71.0
  Participant 2 baseline: number analyzed (Participants) | 2
  Participant 2 baseline | 76.8
  Participant 2 pretest: number analyzed (Participants) | 2
  Participant 2 pretest | 54.8
  participant 2 post tracing: number analyzed (Participants) | 2
  participant 2 post tracing | 51.0
  Participant 2 post games: number analyzed (Participants) | 2
  Participant 2 post games | 94.3
  Participant 3 baseline: number analyzed (Participants) | 3
  Participant 3 baseline | 68.7
  Participant 3 pre test: number analyzed (Participants) | 3
  Participant 3 pre test | 79.9
  Participant 3 post tracing: number analyzed (Participants) | 3
  Participant 3 post tracing | 95.5
  Participating 3 post games: number analyzed (Participants) | 3
  Participating 3 post games | 95.1
  Participant 4 baseline | 44
  Participant 4 pre test | 30.5
  Participant 4 post tracing | 65.8
  Participant 4 post games | 62.3

2. Secondary Outcome: Stylus to Eclipse Area
Time Frame: Base line, Pre and Post training (approximately 3 months)
Population: as for outcome 1
Measure: Number; unit: Degree
Groups:
- SLO Measurements Pre and Post-training: All subjects trained on two computer-based training modules. SLO assessment of changes in fine manual task performance and in retinal functional geography was done before training and after each training module
  SLO measurements pre and post-training
Arm/Group | SLO Measurements Pre and Post-training
Number analyzed (Participants) | 4
Degree
  Participant 1 baseline: number analyzed (Participants) | 1
  Participant 1 baseline | 45.2
  Participant 1 pre test: number analyzed (Participants) | 1
  Participant 1 pre test | 77.6
  Participant 1 post tracing: number analyzed (Participants) | 1
  Participant 1 post tracing | 39.4
  Participant 1 post games: number analyzed (Participants) | 1
  Participant 1 post games | 40.8
  Participant 2 base line: number analyzed (Participants) | 2
  Participant 2 base line | 26.8
  Participant 2 pre test: number analyzed (Participants) | 2
  Participant 2 pre test | 22.6
  Participant 2 post tracing: number analyzed (Participants) | 2
  Participant 2 post tracing | 20.9
  Participant 2 post games: number analyzed (Participants) | 2
  Participant 2 post games | 11.1
  Participant 3 base line: number analyzed (Participants) | 3
  Participant 3 base line | 25
  Participant 3 pre test: number analyzed (Participants) | 3
  Participant 3 pre test | 21.8
  Participant 3 post tracing: number analyzed (Participants) | 3
  Participant 3 post tracing | 47.4
  Participating 3 post games: number analyzed (Participants) | 3
  Participating 3 post games | 47.1
  Participnat 4 base line | 28.4
  Participant 4 pre test | 14.6
  Participant 4 post tracing | 17.8
  Participant 4 post games | 11.8

ADVERSE EVENTS:
Groups:
- Subjects With Bilateral AMD, no Foveal Vision and 20/60 Vision: Crossover design. All subjects undergo all treatments.
  Practice tracing objects and printing with a stylus on a tablet computer: Subjects will have three training modules on a tablet computer: scotoma awareness, line and curve tracing, and video games. The order of modules will be different for different groups of subjects. Training on a module will cease when the subject reaches a performance criterion. Retinal assessments will occur after each training module completion.
Arm/Group | Subjects With Bilateral AMD, no Foveal Vision and 20/60 Vision
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes